CLINICAL TRIAL: NCT02758132
Title: Denosumab Plus Enzalutamide, Abiraterone and Prednisone Compared to Denosumab Plus Enzalutamide Alone for Men With Castrate Resistant Prostate Cancer (CRPC) With Bone Metastases: Clinical Testing and Feasibility of a Serum-based Metabolomics Profile
Brief Title: Denosumab Plus Enzalutamide, Abiraterone and Prednisone Compared to Denosumab Plus Enzalutamide Alone for Men With Castrate Resistant Prostate Cancer (CRPC) With Bone Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accruals
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rosser 2015-1
Record Dates: First submitted 2016-04-11; First posted 2016-05-02 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Castrate-resistant prostate cancer with bone metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Denosumab; enzalutamide; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alliance A031201 (Active Comparator): Denosumab plus enzalutamide, abiraterone and prednisone
  Interventions: Biological: Denosumab; Drug: Enzalutamide; Drug: Abiraterone; Drug: Prednisone
- Standard of Care (Active Comparator): Denosumab plus enzalutamide alone
  Interventions: Biological: Denosumab; Drug: Enzalutamide

INTERVENTIONS:
Biological: Denosumab — One 120 mg subcutaneous injection every four weeks. Protocol therapy will consist of 28-day cycles until no clinical benefit, confirmed disease progression or unacceptable toxicity.
Drug: Enzalutamide — 160 mg enzalutamide by mouth daily
Drug: Abiraterone — 1000 mg abiraterone by mouth daily
  Arms: Alliance A031201
Drug: Prednisone — 5 mg prednisone by mouth twice daily
  Arms: Alliance A031201

SUMMARY:
This is a correlative study to characterize serum metabolites associated with bone deposition, growth and turnover in patients with newly diagnosed metastatic CRPC who are not currently receiving bone targeting agents.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of adenocarcinoma of the prostate with clinical evidence of metastatic disease to the bone.
* Castrate resistant progression of prostate carcinoma, as shown by:

  * Serum testosterone level <50 ng/dL or prior bilateral orchiectomy. Treatment to maintain castrate levels of testosterone should continue, and

    * Either symptomatic progression, or, if patient is asymptomatic then a rising serum PSA in two occasions at least 1 week apart, with minimum pre-treatment serum PSA of 5 ng/dL.
* Patients with nodal disease are eligible.
* Bi-dimensionally measurable disease within the bone.
* Life expectancy of at least 12 weeks.
* ECOG Performance status < 2
* Adequate:

  * Bone marrow function; absolute neutrophil count > 1,500 mm3, platelet count of > 100,000 mm3 and hemoglobin > 9.0 gm/dl.
  * Hepatic function; SGOT/SGPT and conjugated bilirubin less than twice the upper limit of normal.
  * Renal function; serum creatinine ≤ 2 mg/dL (or, if creatinine > 2 mg/dL, then a creatinine clearance of at least 35 ml/min (measured or estimated by the Cockroft formula:

CLcr = [(140-age) x wt (kg)]/[72 x serum creatinine (mg/dL)].

* No evidence of coagulopathy as indicated by PT < 1.5X upper limit of normal.
* Serum calcium (corrected) from 8 to11.5 mg/dL (2 to 2.9 mmol/L) - Patients must sign an informed consent indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

* Patients with variant histologies (e.g., ductal or small cell carcinoma).
* Patients with visceral disease are ineligible.
* Patients who have had prior Sipuleucel-T, docetaxel, cabazitaxel, abiraterone or enzalutamide as a single agent, or in combination therapy.
* Concurrent cancer chemotherapy, radiotherapy or surgery.
* Concurrent serious infection.
* Life threatening illness (e.g., congestive heart failure, uncontrolled angina or myocardial infarction in the prior six months).
* Hypertension uncontrolled by medication.
* Patients who are known to require invasive dental procedures.
* No known or suspected brain metastases (NOTE: patients with treated epidural disease are allowed)
* Administration of any investigational drug within 28 days prior to receipt of denosumab.
* Age ≤ 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alliance A031201 | Standard of Care
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patient expired before completing study
Groups:
- Total: Total of all reporting groups
Arm/Group | Alliance A031201 | Standard of Care | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure Change in Serum-based Metabolites Associated With Bone Deposition, Growth and Turnover in Patients Who Have CRPC With Clinical Evidence of Metastatic Disease to the Bone, All Using Gas Chromatography-time-of-flight Mass Spectrometry (GC-TOFMS).
Time Frame: Prior to Registration, Registration, Day 1 of cycle 4 and 13
Population: Patient expired before completing study
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Measure Time (Months) to Skeletal Related Event (SRE) of Patients on Therapy
Time Frame: Day 1 of each S.O.C cycle (28 days), and until confirmed radiographic disease progression AND initiation of other standard OR investigational agents for prostate cancer, up to 5 years post treatment
Population: Patient expired before completing study
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measure Time (Months) to Progression-free Survival of Patients on Therapy
Time Frame: as for outcome 2
Population: Patient expired before completing study
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measure Time (Months) to Duration of Response of Patients on Therapy.
Time Frame: as for outcome 2
Population: Patient expired before completing study
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Measure Change in Technetium Bone Scintigraphy on Therapy Via Technetium Bone Scintigraphy or Sodium Fluoride (NaF) PET/CT Imaging
Time Frame: Prior to Registration, Day 1 of cycle 4 and 13, Post-Treatment Follow-up (up to 5 years post treatment)
Population: one subject enrolled and they discontinued early from trial, no analysis conducted
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Measure Change in Treatment Response Via RECIST Criteria
Time Frame: as for outcome 2
Population: one subject enrolled and they discontinued early from trial, no analysis conducted
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Evaluate the Effect of Therapy on Quality of Life (QoL) in Patients Via QoL Questionnaire.
Time Frame: Prior to Registration, Registration, Day 1 of cycle 4 and 13
Population: one subject enrolled and they discontinued early from trial, no analysis conducted
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Evaluate the Effect of Therapy on Narcotic Use in Patients on Therapy Via Case Report Forms.
Time Frame: Prior to Registration, Registration, Day 1 of cycle 4 and 13
Population: one subject enrolled and they discontinued early from trial, no analysis conducted
Arm/Group | Alliance A031201 | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were captured over 6 months
Description: adverse event collection performed by standard collection practices, medical chart review, disclosure from subject
Arm/Group | Alliance A031201 | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alliance A031201 (N=0) | Standard of Care (N=1)
intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) — subject was admitted to the hospital on 9/3/2016. Subject had a significant history of CVA (stroke) with atrial fibrillation. Patient elected hospice and care expired on 9/8/2016. The event was a grade 5 and deemed unrelated to study treatment.

LIMITATIONS AND CAVEATS:
Trial was terminated early due to low accrual of one subject. Data analysis not conducted due to the one enrolled subject not receiving all the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes